CLINICAL TRIAL: NCT02385058
Title: Double-Blind, Placebo-Controlled, Randomized, Prospective, Two-Stage, Two-Arm Study to Evaluate the Efficaciousness and Safety of a Double Treatment Plan Using a Combination of Mebendazole and Quinfamide for Treating Intestinal Helminthiasis and Amebiasis in the Mexican Population
Brief Title: Study to Evaluate Efficacy and Safety of a Double Treatment Plan Using a Combination of Mebendazole and Quinfamide for Treating Intestinal Helminthiasis and Amebiasis in the Mexican Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003685; JC/AMO/REC/0605 (Other: Janssen-Cilag Ltd); MEBENDAZOLGAI3001 (Other: Janssen-Cilag Ltd)
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Helminthiasis; Amoebiasis
Keywords: Helminthiasis; Amoebiasis; Mebendazole; Quinfamide; Mexican population
MeSH Terms: conditions — Helminthiasis; Amebiasis | interventions — Mebendazole; quinfamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mebendazole + Quinfamide (Experimental): Participants will receive mebendazole 600 milligram (mg) and quinfamide 200 mg tablets orally once starting on Day 1 and 21 in both Phase 1 and 2.
  Interventions: Drug: Mebendazole; Drug: Quinfamide
- Mebendazole + Quinfamide + Placebo (Experimental): Participants will receive mebendazole 600 mg and quinfamide 200 mg tablets orally once starting on Day 1 in Phase 1 and placebo tablets orally once starting on Day 21 in Phase 2.
  Interventions: Drug: Mebendazole; Drug: Quinfamide; Drug: Placebo

INTERVENTIONS:
Drug: Mebendazole — Mebendazole 600 milligram (mg) tablet orally once starting on Day 1 and 21.
Drug: Quinfamide — Quinfamide 200 mg tablet orally once starting on Day 1 and 21.
Drug: Placebo — Placebo tablet orally once starting on Day 21.
  Arms: Mebendazole + Quinfamide + Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of the combination of mebendazole plus quinfamide for the treatment of intestinal helminthiasis and amoebiasis in Mexican population.

DETAILED DESCRIPTION:
This is a double-blind (neither investigator nor participant knows which treatment the participant receives), placebo-controlled (placebo is an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial), randomized (study medication assigned to participants by chance), prospective (study following patients forward in time) study. The total study duration for each participant will be approximately 48 days. The study will consist of 3 parts: Screening Phase (5 days) and double-blind treatment Phase (from Day 1 to 21, consists of Phase-1 and Phase-2) and follow-up Phase (from Day 21 to 43). Participants will receive mebendazole (600 milligram [mg]) and quinfamide (200 mg) tablets orally once starting on Day 1 and mebendazole 600 mg and quinfamide (200 mg) or placebo tablets orally once starting on Day 21. Efficacy will be primarily evaluated by percentage of participants with eradication of helminthic and/or protozoa. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Minors whose parents or tutor grant his/her informed consent in writing to participate in the study. Adult participants that give their informed consent in writing to participate
* Participants having a copro-parasitoscopy test (scatology) (at least 1 with a series of 3) qualitative and quantitative and/or search of live amoeba, that comes out positive for one or more of the following parasites: Ascaris lumbricoides, Enterobius vermicularis, Trichuris trichuria, Taenia solium, Necator americanus, Ancylostoma duodenale and Trophozoites of Entamoeba histolytica
* With at least two or more of the following symptoms: Anorexia, Nausea, Vomit, Abdominal pain, Diarrhea, Constipation, Evacuations with mucus, Evacuations with blood, Gas discharge, Weight loss and Bruxism

Exclusion Criteria:

* Participants with any known allergy to any of the drugs used in the investigation
* Female Participant in reproductive age not using an adequate contraceptive method
* Pregnant or lactating Participant
* Participant with any life-threatening condition (cancer, AIDS, etc.)
* Participant known to be a carrier of some illness that alters the metabolism or drug excretion (hepatic or renal illness) interfering with the absorption (malabsorption) or interferes with the evaluation of the Participant during the study
* Participants that have taken any antiparasitic drug 14 days previous to his/her inclusion in this clinical investigation protocol
* Participants with diagnosis of extra-intestinal amoebiasis

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-10; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Eradication of Helminthic and/or Protozoa (Trophozoites of Amoeba) | Day 21
  Participants must show the results of a negative copro-parasitoscopy exam and fresh amoeba test after the first and second treatment phase. Those participants presenting a positive result during the control exams will be considered as "Therapeutic failure".
Percentage of Participants with Eradication of Helminthic and/or Protozoa (Trophozoites of Amoeba) | Day 43
  Participants must show the results of a negative copro-parasitoscopy exam and fresh amoeba test after the first and second treatment phase. Those participants presenting a positive result during the control exams will be considered as "Therapeutic failure".

SECONDARY OUTCOMES:
Percentage of Participants with Abdominal Symptoms Relieve | Day 43
  Evaluation of abdominal symptoms relief will be carried by the questionnaires, each one of the symptoms presence will be evaluated determining its presence or absence, intensity, and changes throughout the treatment period.
Percentage of Participants with Improved Quality of Life | Day 43
  Evaluation of improved quality of life will be carried by the questionnaires, the results will be evaluated according to the symptomatic satisfaction scales, scale ranges from Excellent to Terrible (Excellent = very satisfied, Good= satisfied, Poor= more or less satisfied, Bad= unsatisfied and Terrible= very unsatisfied), which should show that there was an improvement in the sensation of wellbeing of the participant compared with the symptoms provoked by the presence of the intestinal parasitosis.
Number of Participants with Adverse Events (AEs) and Serious AEs | Screening up to follow-up (Day 43)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (1):
- Mexico City, Mexico